CLINICAL TRIAL: NCT01447511
Title: Pharmacogenetics of Warfarin Induction and Inhibition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Collaborators: National Institute of General Medical Sciences (NIGMS) (NIH)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 0807M38361; P01GM032165-26 (NIH)
Record Dates: First submitted 2010-01-29; First posted 2011-10-06 (Estimated); Results first posted 2014-08-18 (Estimated); Last update posted 2018-11-14 (Actual); Status verified 2018-10

CONDITIONS: Healthy
Keywords: Drug Interactions; Warfarin; Genetics; CYP2C9; Healthy Volunteers
MeSH Terms: interventions — Warfarin; Fluconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (5):
- CYP2C9*1/*1 Genotype (Other): This genotype is considered the wild type genotype. Individuals with the CYP2C9*1/*1 genotype have two *1 alleles and participated in the following interventions: Control - Warfarin only, Fluconazole - Warfarin, and Rifampin - Warfarin.
  Interventions: Drug: Control - Warfarin only; Drug: Fluconazole - Warfarin; Drug: Rifampin - Warfarin
- CYP2C9*1B/*1B Haplotype (Other): Individuals with the CYP2C9*1B/*1B haplotype have two CYP2C9*1B alleles and participated in the following interventions: Control - Warfarin only and Rifampin - Warfarin.
  Interventions: Drug: Control - Warfarin only; Drug: Rifampin - Warfarin
- CYP2C9*1/*3 Genotype (Other): Individuals with the CYP2C9*1/*3 genotype have one *1 allele and one *3 allele and participated in the following interventions: Control - Warfarin only, Fluconazole - Warfarin, and Rifampin - Warfarin.
  Interventions: Drug: Control - Warfarin only; Drug: Fluconazole - Warfarin; Drug: Rifampin - Warfarin
- CYP2C9*2/*3 Genotype (Other): Individuals with the CYP2C9*2/*3 genotype have one *2 and one *3 allele and participated in the following interventions: Control - Warfarin only, Fluconazole - Warfarin, and Rifampin - Warfarin.
  Interventions: Drug: Control - Warfarin only; Drug: Fluconazole - Warfarin; Drug: Rifampin - Warfarin
- CYP2C9*3/*3 Genotype (Other): Individuals with the CYP2C9*3/*3 genotype have two *3 alleles and participated in the following interventions: Control - Warfarin only, Fluconazole - Warfarin, and Rifampin - Warfarin.
  Interventions: Drug: Control - Warfarin only; Drug: Fluconazole - Warfarin; Drug: Rifampin - Warfarin

INTERVENTIONS:
Drug: Control - Warfarin only — A single 10 mg warfarin dose taken at the start of the study period. No other medications taken during this study period.
  Other Names: Coumadin
Drug: Fluconazole - Warfarin — A single 10 mg warfarin dose taken at the start of the study period. 400 mg fluconazole taken every morning starting a week before the start of the study period and continuing throughout the study period.
  Other Names: Diflucan; Coumadin
  Arms: CYP2C9*1/*1 Genotype; CYP2C9*1/*3 Genotype; CYP2C9*2/*3 Genotype; CYP2C9*3/*3 Genotype
Drug: Rifampin - Warfarin — A single 10 mg warfarin dose taken at the start of the study period. 300 mg rifampin taken every morning starting a week before the start of the study period and continuing throughout the study period.
  Other Names: Rifadin; Coumadin

SUMMARY:
This research study will help determine how a person's genetic makeup affects their response to drugs, the ability of the body to break down drugs, and their potential to experience an interaction between drugs. The investigators are investigating the drug interactions with the commonly used anticoagulant drug called warfarin. Warfarin is used for the treatment and prevention of life-threatening abnormal blood clots such as deep vein thrombosis, heart attacks, and strokes. The investigators chose warfarin for this study because it is a commonly used drug and must be monitored closely to avoid side effects. The investigators are interested in studying whether individuals with certain genetic profiles react differently to warfarin when it is combined with other drugs. This research is being done to see if certain genetic profiles require us to adjust warfarin doses differently than is needed for the general population. Genetic profiles of subjects are determined from their participation in the Pharmacogenetics Registry study (investigator Richard Brundage, University of Minnesota).

The study hypothesis is: Functionally defective CYP2C9 alleles attenuate the warfarin-fluconazole inhibitory interaction and exacerbate the warfarin-rifampin inductive interaction.

DETAILED DESCRIPTION:
The research question is: How does CYP2C9 genotype modify warfarin drug interactions?

People differ in their genetic makeup. This includes differences in genes involved in drug metabolism, transport, and effect in the body. People with certain genetic profiles produce altered enzymes, transporters, and receptors that may respond in different ways to drugs. Altered enzymes cause some drugs to be broken down at a different rate than normal. As a result, drug concentrations build up in the blood, and increase the risk of side effects. Furthermore, when two drugs are taken together, the possibility exists for the drugs to interact, with one drug causing a change in the metabolism of the other or both of the drugs. It is not known whether people with an altered genetic makeup also have an altered experience with drug interactions. Altered drug transporters can affect the absorption and elimination of drugs as compared to normal causing differences in how long the drug stays in the body. Finally, altered drug receptors can respond differently to drugs and, thus, produce altered desired or undesired effects.

In this study, the investigators will be investigating the drug interactions with the commonly used anticoagulant drug warfarin in subjects with five different CYP2C9 genotypes. The CYP2C9 genotype is particularly important because this drug metabolizing enzyme governs the metabolic clearance of the more potent chemical entity (the S-enantiomer) of the drug. Warfarin is used for the treatment and prevention of life-threatening abnormal blood clots such as deep vein thrombosis, myocardial infarction, and strokes. The investigators chose warfarin for this study because it is a commonly used drug and must be monitored closely to avoid side effects. The investigators are interested in studying whether individuals with certain genetic alleles of the CYP2C9 genotype react differently to warfarin when it is combined with an antifungal (fluconazole) that inhibits CYP2C9-mediated metabolism and an antibiotic (rifampin) that induces CYP2C9-mediated metabolism. This research is being done to see if certain genetic profiles require us to adjust warfarin doses differently than is needed for the general population.

The study hypothesis is: Functionally defective CYP2C9 alleles attenuate the warfarin-fluconazole inhibitory interaction and exacerbate the warfarin-rifampin inductive interaction.

ELIGIBILITY:
Inclusion Criteria:

* Subjects will be 18-60 years old.
* Women of child bearing age must be willing to use measures to avoid conception during the study period.
* Subjects must agree not to take any known substrates, inhibitors, inducers or activators of either CYP2C9 or CYP3A4 from 1 week prior to the start of each study through the last day of study.

Exclusion Criteria:

* Current cigarette smoker
* Abnormal renal, liver function tests, physical exam, or recent history of hepatic, renal, gastrointestinal or neoplastic disease.
* Allergy to warfarin, fluconazole or rifampin and other chemically related drugs.
* Recent ingestion (< 1 week) of any medication known to be metabolized by or alter CYP2C9 or CYP3A4 activity.
* A positive pregnancy test at the time of the pharmacokinetic study.
* Lab tests indicative of abnormal blood clotting capacity.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 39 (Actual)
Dates: Start 2009-05; Primary Completion 2013-06 (Actual); Study Completion 2013-06 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Richard Brundage, PhD, Principal Investigator — University of Minnesota
Locations (1):
- Clinical and Translational Science Institute, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Flora DR, Rettie AE, Brundage RC, Tracy TS. CYP2C9 Genotype-Dependent Warfarin Pharmacokinetics: Impact of CYP2C9 Genotype on R- and S-Warfarin and Their Oxidative Metabolites. J Clin Pharmacol. 2017 Mar;57(3):382-393. doi: 10.1002/jcph.813. Epub 2016 Sep 22. PMID 27539372

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: Thirty-nine participants were enrolled in the study; however, only twenty-nine of the enrolled participants participated in the study. Per study protocol, participants with the CYP2C9*1B/*1B haplotype did not complete the Fluconazole Period. Individuals with the CYP2C9*1B/*1B haplotype only completed the Control Period and Rifampin Period.
Groups:
- CYP2C9*1/*1 Genotype: This genotype is considered the wild type genotype. Individuals with the CYP2C9*1/*1 genotype have two *1 alleles and participated in the following periods: Control Period, Fluconazole Period, and Rifampin Period.
- CYP2C9*1B/*1B Haplotype: Individuals with the CYP2C9*1B/*1B haplotype have two *1B alleles and participated in the following periods: Control Period and Rifampin Period.
- CYP2C9*1/*3 Genotype: Individuals with the CYP2C9*1/*3 genotype have one *1 allele and one *3 allele and participated in the following periods: Control Period, Fluconazole Period, and Rifampin Period.
- CYP2C9*2/*3 Genotype: Individuals with the CYP2C9*2/*3 genotype have one *2 allele and one *3 allele and participated in the following periods: Control Period, Fluconazole Period, and Rifampin Period.
- CYP2C9*3/*3 Genotype: Individuals with the CYP2C9*3/*3 genotype have two *3 alleles and participated in the following periods: Control Period, Fluconazole Period, and Rifampin Period.
Period: Control Period
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype
Started | 8 | 5 | 9 | 3 | 4
Completed | 8 | 5 | 9 | 3 | 4
Not Completed | 0 | 0 | 0 | 0 | 0
Period: Fluconazole Period
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype
Started | 8 | 0 | 9 | 3 | 4
Completed | 8 | 0 | 8 | 3 | 4
Not Completed | 0 | 0 | 1 | 0 | 0
Period: Rifampin Period
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype
Started | 8 | 5 | 8 | 3 | 4
Completed | 8 | 5 | 8 | 2 | 4
Not Completed | 0 | 0 | 0 | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype | Total
Number analyzed (Participants) | 8 | 5 | 9 | 3 | 4 | 29
Age, Continuous [Median (Full Range); unit: years] | 22 [19 to 54] | 23 [22 to 31] | 26 [18 to 52] | 28 [21 to 51] | 29 [19 to 33] | 25 [18 to 54]
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 1 | 0 | 0 | 1
  Between 18 and 65 years | 8 | 5 | 8 | 3 | 4 | 28
  >=65 years | 0 | 0 | 0 | 0 | 0 | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 2 | 5 | 3 | 0 | 14
  Male | 4 | 3 | 4 | 0 | 4 | 15
Region of Enrollment [Number; unit: participants]
  United States | 8 | 5 | 9 | 3 | 4 | 29

OUTCOME MEASURES:

1. Primary Outcome: Warfarin Clearance.
Description: Warfarin enantiomer (S-warfarin and R-warfarin) clearance was measured in healthy volunteers genotyped for CYP2C9*1/*1, CYP2C9*1B/*1B, CYP2C9*1/*3, CYP2C9*2/*3 and CYP2C9*3/*3 to determine the magnitude of the warfarin-fluconazole (inhibition) and warfarin-rifampin (induction) drug interactions.
Time Frame: Over three (two for CYP2C9*1B/*1B participants) 12-16 day study periods.
Population: Participants with the CYP2C9*1B/*1B haplotype did not participate in the fluconazole period (inhibition). One CYP2C9*1/*3 participant only completed the control period. One CYP2C9*2/*3 participant only completed the control and fluconazole (inhibition) study periods.
Measure: Mean (Standard Deviation); unit: mL/h
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype
Number analyzed (Participants) | 8 | 5 | 9 | 3 | 4
mL/h
  S warfarin - Control Period | 282 (62) | 246 (69) | 180 (49) | 84 (7) | 71 (5)
  R warfarin - Control Period | 136 (37) | 124 (54) | 122 (27) | 95 (10) | 153 (38)
  S warfarin - Fluconazole Period | 89 (17) | NA (NA) — Participants with the CYP2C9*1B/*1B haplotype did not participate in the fluconazole period per study protocol. | 68 (22) | 35 (7) | 36 (6)
  R warfarin - Fluconazole Period | 66 (13) | NA (NA) — Participants with the CYP2C9*1B/*1B haplotype did not participate in the fluconazole period per study protocol. | 68 (10) | 55 (13) | 72 (7)
  S warfarin - Rifampin Period | 520 (69) | 486 (151) | 347 (140) | 195 (20) | 157 (8)
  R warfarin - Rifampin Period | 342 (64) | 307 (151) | 339 (64) | 368 (74) | 406 (108)
Statistical Analysis 1: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean S-warfarin clearance among the five CYP2C9 genotypes under control conditions is the same; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 2: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean S-warfarin clearance among the five CYP2C9 genotypes under fluconazole conditions is the same; Test type: Superiority or Other; p = 0.0001, ANOVA
Statistical Analysis 3: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean S-warfarin clearance among the five CYP2C9 genotypes under rifampin conditions is the same; Test type: Superiority or Other; p < 0.0001, ANOVA
Statistical Analysis 4: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean R-warfarin clearance among the five CYP2C9 genotypes under control conditions is the same; Test type: Superiority or Other; p = 0.3058, ANOVA
Statistical Analysis 5: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean R-warfarin clearance among the five CYP2C9 genotypes under fluconazole conditions is the same; Test type: Superiority or Other; p = 0.3278, ANOVA
Statistical Analysis 6: Comparison: CYP2C9*1/*1 Genotype vs CYP2C9*1B/*1B Haplotype vs CYP2C9*1/*3 Genotype vs CYP2C9*2/*3 Genotype vs CYP2C9*3/*3 Genotype; The null hypothesis is that the mean R-warfarin clearance among the five CYP2C9 genotypes under rifampin conditions is the same; Test type: Superiority or Other; p = 0.6155, ANOVA

ADVERSE EVENTS:
Arm/Group | CYP2C9*1/*1 Genotype | CYP2C9*1B/*1B Haplotype | CYP2C9*1/*3 Genotype | CYP2C9*2/*3 Genotype | CYP2C9*3/*3 Genotype
Serious Adverse Events (participants affected / at risk) | 0/8 | 0/5 | 0/9 | 0/3 | 0/4
Other Adverse Events (participants affected / at risk) | 4/8 | 4/5 | 6/9 | 0/3 | 2/4
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | CYP2C9*1/*1 Genotype (N=8) | CYP2C9*1B/*1B Haplotype (N=5) | CYP2C9*1/*3 Genotype (N=9) | CYP2C9*2/*3 Genotype (N=3) | CYP2C9*3/*3 Genotype (N=4)
Blood in Bowel (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Body Ache (General disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 1 (2) | 0 (0) | 0 (0)
Chills (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Common Cold Symptoms (General disorders) | 0 (0) | 0 (0) | 4 (7) | 0 (0) | 1 (1)
Diarrhea (Gastrointestinal disorders) | 1 (1) | 1 (1) | 1 (1) | 0 (0) | 0 (0)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 2 (2) | 0 (0) | 1 (1)
Dry Lips (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Fatigue (General disorders) | 0 (0) | 3 (4) | 2 (2) | 0 (0) | 0 (0)
Fever (General disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Headache (Nervous system disorders) | 0 (0) | 2 (5) | 4 (4) | 0 (0) | 1 (1)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 2 (4) | 0 (0) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0)
Skin Abrasion (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Stomach Pain (Gastrointestinal disorders) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes